CLINICAL TRIAL: NCT01569308
Title: Pulse Pressure Variation Helps to Predict Fluid Responsiveness in Patients Ventilated With Low Tidal Volumes
Status: Completed | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: 06-109
Record Dates: First submitted 2012-03-14; First posted 2012-04-03 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Hemodynamic Instability
Keywords: Cardiac output; Pulse pressure variation; Fluid responsiveness; Low tidal volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Objective: To determine the value of pulse pressure variation (ΔRESPPP) to predict fluid responsiveness in patients ventilated with low tidal volumes (VT), and to investigate whether a lower ΔRESPPP cut-off point should be used when patients are ventilated with low tidal volumes.

Methods: This cross-sectional, observational study included 37 critically ill patients with acute circulatory failure requiring fluid challenge. They were sedated and mechanically ventilated with Tidal Volume (VT) 6-7 ml/kg IBW (ideal body weight), monitored by pulmonary artery catheter and arterial line. Mechanical ventilation and hemodynamic parameters, including ΔRESPPP, were measured before and after fluid challenge with 1,000 ml crystalloids or 500 ml colloids. Fluid responsiveness was defined as an increase of at least 15% in cardiac index.

The present study was designed to (1) determine the value of ΔRESPPP to predict fluid responsiveness in patients ventilated with low tidal volumes, and (2) to investigate whether a lower ΔRESPPP cut-off point should be used when patients are ventilated with low tidal volumes.

The study hypothesis is not a good predictor of fluid responsiveness in patients ventilated with low tidal volumes.

DETAILED DESCRIPTION:
Volume expansion is frequently used to treat critically ill patients with acute circulatory failure. The goal of volume expansion is to increase left ventricular stroke volume and consequently cardiac output. However, about 50% of patients with acute circulatory failure will respond to fluid challenge (preload- dependent patients). Therefore, the ability to predict fluid responsiveness in critically ill patients is crucial, particularly for ARDS patients because of increased alveolar-capillary membrane permeability, and avoiding unnecessary fluid loading has been shown to have a positive effect on patient outcome.Among the dynamic parameters used at the bedside to identify fluid responsiveness, pulse pressure variation (ΔRESPPP) is one of the most accurate in patients with acute circulatory failure receiving invasive mechanical ventilation. However, most studies evaluated patients ventilated with large tidal volumes (≥ 8 ml/kg). Therefore, the validity of ΔRESPPP to identify fluid responsiveness is still debated when lower tidal volumes are used.

The current literature about its performance during ventilation with low tidal volumes is unclear, and opposite conclusions have been drawn. The present study was designed to (1) determine the value of ΔRESPPP to predict fluid responsiveness in patients ventilated with low tidal volumes, and (2) to investigate whether a lower ΔRESPPP cut-off point should be used when patients are ventilated with low tidal volumes.

Methods: This cross-sectional, observational study included 37 critically ill patients with acute circulatory failure requiring fluid challenge. They were sedated and mechanically ventilated with Tidal Volume (VT) 6-7 ml/kg IBW (ideal body weight), monitored by pulmonary artery catheter and arterial line. Mechanical ventilation and hemodynamic parameters, including ΔRESPPP, were measured before and after fluid challenge with 1,000 ml crystalloids or 500 ml colloids. Fluid responsiveness was defined as an increase of at least 15% in cardiac index.

Patients were followed for 28 days or until discharge from the ICU.

Study Protocol Patients were sedated with midazolan and fentanyl (score of -4 to -5 in the Richmond Agitation Sedation Scale)and ventilated in controlled pressure or controlled volume mode (Servo I system v.12 or Servo 900 C, Siemens, Sweden) with VT < 8 ml/kg IBW (51 + 0.9[height in cm- 152.9] for men and 45.5 + 0.91[height in cm- 152.9] for women). Ventilatory and hemodynamic variables were measured before and after FC with the patients in a supine position. Zero pressure was measured at the midaxillary line. The correct position of the pulmonary artery catheter in West's zone 3 was checked as described in the literature.

Fluid challenge was performed with 1000 ml 0.9% saline solution or lactated Ringer's solution (n=36) or 500 ml hydroxy-ethyl-starch solution 6% 130/0.4 for 30 minutes (n=2).

Hemodynamic Parameters

Variations in arterial pulse pressure were visualized on bedside monitors (HP S66 and PHILIPS IntelliVue, MP60, Germany) and measured with the cursor for each of 5 breathing cycles. ΔRESPPP was calculated using the following equation:

ΔRESPPP (%) = 100 x (PPmax - PPmin) / [(PPmax + PPmin)/2]

where PPmax and PPmin are the maximal pulse pressure at inspiration and the pulse pressure obtained on expiration, respectively.

A pulmonary artery catheter (Edwards Healthcare, Irvine, CA) was used to measure cardiac output according to the thermal dilution method (3 injections of 10ml 0.9% saline solution), systolic, diastolic and mean pulmonary arterial pressures, pulmonary artery occlusion pressure (PAOP, mmHg), central venous pressure (CVP, mmHg), and mixed venous saturation (SvO2). Mean arterial pressure (MAP, mmHg), measured using the arterial line, and heart rate (HR, bpm) were also recorded. All measurements were made at the end of expiration, before and after FC. Patients were defined as fluid responders when cardiac index increased at least 15% of baseline value.

Ventilation Parameters The following ventilatory parameters were measured: inspiratory and expiratory tidal volume, respiratory rate (RR), plateau pressure (cmH2O), peak pressure (cmH2O), total positive end-expiratory pressure (PEEPtot), static compliance (Cst) and driving pressure (DP= Pplat-PEEP). All measurements were made before and after FC.

Statistical Analysis Sample size was defined as 38 patients for estimation of the correlation between CI and ΔRESPPP 0.5 (moderate to high magnitude), with a level of significance of 0.05 and power of 90%.

The effects of FC on hemodynamic parameters were assessed using a paired Student's t-test for normally distributed variables or a nonparametric Wilcoxon Signed Rank test for non-normally distributed variables. The comparison of hemodynamic parameters between both groups at baseline and after FC was assessed using a two sample Student's t-test or a nonparametric Mann-Whitney U test. Results were expressed as mean values±SD or median (25-75 percentiles).

Receiver operating characteristic (ROC) curves were constructed to evaluate the ability of ΔRESPPP, ΔRESPPP/DP, CVP and PAOP to predict fluid responsiveness. The best cut-off value for ΔRESPPP ROC curve was determined for the entire population. In addition, measures of diagnostic performance were calculated: sensitivity, specificity, predictive values and likelihood ratio. Linear correlations were tested using the Spearman rank method. Data were analyzed using SPSS 15.0. A p value <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years
* Hemodynamic instability defined as need for norepinephrine infusion and/or intravascular fluid administration to maintain systolic arterial blood pressure > 90 mm Hg
* Arterial line in place (radial or femoral)
* Pulmonary arterial catheter in place

Exclusion Criteria:

* Presence of cardiac arrhythmias
* Presence of pneumothorax
* Presence of heart valve disease or intracardiac shunt
* Previously diagnosed right ventricular insufficiency

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients age ≥ 16 years, from both genders, admitted to the HCPA ICU, receiving invasive mechanical ventilation, with hemodynamic instability defined as need for norepinephrine infusion and/or intravascular fluid administration to maintain systolic arterial blood pressure > 90 mm Hg; with arterial line in place (radial or femoral) and pulmonary arterial catheter in place.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2006-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Increase in cardiac index at least 15% of baseline value. | Cardiac index was measured at the end of a 30 minutes fluid challenge.
  Patients were sedated and ventilated in controlled pressure or controlled volume mode (Servo I system v.12 or Servo 900 C, Siemens, Sweden) with VT < 8 ml/kg ideal body weight. Ventilatory and hemodynamic variables were measured before and after FC with the patients in a supine position. Fluid challenge was performed with 1000 ml 0.9% saline solution or lactated Ringer's solution or 500 ml hydroxy-ethyl-starch solution 6% 130/0.4 for 30 minutes. The increase in cardiac index was measured immediately after fluid challenge.

SECONDARY OUTCOMES:
Mortality | 28 days
  Patients were followed for 28 days or until ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto Friedman, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Oliveira-Costa CD, Friedman G, Vieira SR, Fialkow L. Pulse pressure variation and prediction of fluid responsiveness in patients ventilated with low tidal volumes. Clinics (Sao Paulo). 2012 Jul;67(7):773-8. doi: 10.6061/clinics/2012(07)12. PMID 22892922